CLINICAL TRIAL: NCT05098080
Title: 2021-PT054: A Randomized Phase I Open-Label, Placebo-Controlled, Dose Escalation Study to Evaluate Safety and Pharmacokinetics of Hutrukin Via Intravenous Administration in Healthy Subjects.
Brief Title: Hutrukin to Analyze Safety and PK in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-PT054
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-12

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Eight healthy subjects will be in each of the three dose cohorts (1,000 mg, 3,000 mg and 5,000 mg). For each dose cohort, six subjects will be administered Hutrukin and two will be administered placebo and the study will not proceed to the next dose level unless the tested dose level has been deemed to have acceptable tolerability and safety. Subjects will undergo blood sampling at multiple time points up to 28 days. Subjects will also be evaluated for the development of anti-drug antibodies (ADA).
  Dose escalation will utilize a 6+2 design with sentinel dosing and doses will be explored in cohort of 8 subjects (6 active drug and 2 placebo). There are two sub-groups, the first is comprised of one subject receiving Hutrukin and one subject receiving placebo, the second sub-group is comprised of five subjects receiving active drug and one subject receiving placebo. A 24-hour observation window will be given before enrolling the subjects in the second sub-group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hutrukin (Active Comparator): At least six healthy subjects in each of the three dose cohorts (1000 mg, 3000 mg, and 5000 mg), will be administered Hutrukin.
  Interventions: Biological: Hutrukin
- Placebo (Placebo Comparator): At least two healthy subjects in each of the three dose cohorts (1000 mg, 3000 mg, and 5000 mg), will be administered placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Hutrukin — Hutrukin that binds the human cytokine IL-1α with high affinity and is an effective blocker of IL-1α biological activity. Hutrukin is a True Human™ therapeutic antibody. That is, the antibody was generated by a natural human immune response and was cloned directly from a human peripheral B lymphocyte. No in vitro affinity maturation or modifications have been made to improve its natural binding affinity. A true human antibody should be effectively non-immunogenic in humans and thus exhibit optimal activity and pharmacokinetics indistinguishable from native IgG1 immunoglobulin.
  Arms: Hutrukin
Biological: Placebo — Placebo control for Hutrukin IV push.
  Arms: Placebo

SUMMARY:
The study will be a Phase I, open label, safety and pharmacokinetics study of HutrukinTM in at least eight healthy subjects in each of the three dose cohorts (1,000 mg, 3,000 mg and 5,000 mg).

DETAILED DESCRIPTION:
Study Title: A Randomized Phase I Open-Label, Placebo-Controlled, Dose Escalation Study to Evaluate Safety and Pharmacokinetics of Hutrukin via Intravenous Administration in Healthy Subjects

Sponsor: XBiotech USA, Inc.

Study Chair: Neha Reshamwala, MD

Number of Planned Subjects: 24 healthy subjects with 8 subjects in each of the dose cohorts of HutrukinTM.

Approximate Duration:

Approximately 38 days which includes a screening period of up to 10 days followed by one intravenous push of Hutrukin and then evaluation over 28 days. Blood will be sampled at various time points for blood chemistry, hematological assessment and Hutrukin serum/plasma concentrations. Safety and tolerability will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 and weight ≥40 kg.
2. Adequate bone marrow function defined as:

   * absolute neutrophil count (neutrophil and bands) of ≥ 1,500/mm3 (≥ 1.5 x 109/L)
   * platelet count > 150,000/mm3
   * hemoglobin of ≥ 10 g/dL
3. Adequate renal function, defined by serum creatinine ≤ 1.5 x lab ULN.
4. Adequate hepatic function defined as:

   * serum albumin ≥ 3.0 g/dL
   * total bilirubin ≤ 1.5 times lab ULN.
   * alanine aminotransferase (ALT) ≤ 2.0 times lab ULN.
   * aspartate aminotransferase (AST) ≤ 2.0 times lab ULN
5. For female subjects of childbearing potential WOCBP, a negative pregnancy test at screening and the female subjects must agree to either abstain from sexual intercourse or use reliable, effective contraception such as hormonal contraceptive, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, or use of a condom by their partner. Women of non-childbearing potential include those who cannot get pregnant medically, including post-menopausal women and those with a history of hysterectomy or surgical sterilization.
6. Male participants must agree to abstain from sexual intercourse or use a reliable, effective contraceptive method, such as condoms, or have had a vasectomy. Alternatively, female partners of male subjects enrolled in the study must use reliable, effective contraception such as hormonal contraceptive, intrauterine device (IUD), diaphragm with spermicide, or contraceptive sponge.
7. Signed and dated Institutional Review Board (IRB) approved informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

1. Treatment with any biologicals (including intravenous immunoglobulin) or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
2. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within the past 6 months.
   * Uncontrolled angina within the past 3 months.
   * Congestive heart failure within the past 3 months, defined as New York Heart Association (NYHA) Class II or higher.
   * Uncontrolled hypertension (blood pressure >160 mm Hg systolic or >100 mm Hg diastolic).
3. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
4. Treatment with immunosuppressant agents, including corticosteroids or cyclosporine within the last 4 weeks.
5. History of any clinically significant medical disorders the investigator decides should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
7. Abnormal ECG with any clinically significant findings or with QTc >470 ms.
8. Serious infection (example: sepsis, pneumonia, or pyelonephritis), or have been hospitalized or received intravenous (IV) antibiotics for a serious infection during the 3 months prior to the screening visit.
9. Infectious disease:

   • Positive HIV, RPR, Hepatitis B or C, TB (QuantiFERON-TB Gold (QFT)/ IGRA)
10. History of immunodeficiency.
11. Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding.
12. Major surgery within 28 days prior to Day 0.
13. History of progressive multifocal leukoencephalopathy (PML) or other demyelinating disease.
14. History of malignancy before screening with the exception of squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment related adverse events assessed according to CTCAE v5.0 of one single intravenous dose of HutrukinTM in healthy subjects at each dose level. | 28 days
  Participants will be monitored for acute reactions, blood chemistry and hematology immediately after dosing and at multiple time points up to 28 days. All adverse events will be documented at multiple time points and assessed in terms those possibly, probably and definitely related to test article according to CTCAE v5.0 criteria. Anti-drug antibodies (ADA) will also be evaluated.

SECONDARY OUTCOMES:
Maximum plasma concentration of test article | 28 days
  The maximum plasma concentration will be assessed using a proprietary immunoassay to detect circulating HutrukinTM.
Plasma concentration at various time points including terminal concentration | 28 days
  Terminal plasma concentration will be assessed at 28 days.
Half-life | 28 days
  Half-life will be assessed.
Total exposure | 28 days
  Area under the curve will be determined based on measured plasma levels over 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Reshamwala, MD, Principal Investigator — BioBehavioral Research of Austin
Locations (1):
- BioBehavioral Research of Austin, A Telemed2U Company, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No It is not yet known if there will be a plan to make IPD available